CLINICAL TRIAL: NCT05057910
Title: Evaluation of SARS-CoV-2 RBD Antibody in Vaccinated Healthcare Workers at My Duc Hospital: a Cross-sectional Study
Brief Title: SARS-CoV-2 (Covid-19) RBD Antibody in My Duc Hospital Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10/21/ĐĐ-BVMĐ
Record Dates: First submitted 2021-09-20; First posted 2021-09-27 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Covid19; Vaccine Reaction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 IgG II Quant — 3ml of blood samples are collected, contained in heparin-free tubes, and centrifuged. Blood serum samples are collected and stored at the -80 Celcius degree. SARS-CoV-2 IgG antibodies in human serum and plasma are detected using chemiluminescent microparticle immunoassay (CMIA) technology on the ARCHITECT I 1000r System. Quality Control procedures will take place once daily, with three levels: one negative control and two positive controls. Sample, SARS-CoV-2 antigen-coated paramagnetic microparticles, and assay diluent are combined and incubated. The SARS-CoV-2 IgG antibodies present in the sample bind to the antigen-coated microparticles. The resulting chemiluminescent reaction is measured as a relative light unit (RLU). There is a direct relationship between the titres of IgG antibodies to SARS-CoV-2 in the sample and the RLU detected by the system optics. Interpretation of Results: < 50.0 AU/mL, Negative, ≥ 50.0 AU/mL, Positive

SUMMARY:
To evaluate the immune response to the ChAdOx1 nCoV-19 vaccine by measuring the titers of antibody against the SARS-CoV-2 spike protein receptor binding domain (RBD) among healthcare workers of My Duc Hospital and investigate potential associations of vaccine protection against infection in this population. The study's data can suggest the groundwork for the development of predictive models for post-vaccination protection in the Vietnamese population as well as for establishing vaccination strategies to control disease outbreaks in the future.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome caused by coronavirus 2 (SARS-CoV-2) emerged in December 2019 from Wuhan, China. This pandemic quickly spread to many countries and became a global health challenge with profound impacts on human health as well as on economic and social life. As of September 12, 2021, according to the statistic registry of the Ministry of Health of Vietnam, the total number of SARS-CoV-2 infections is 624,547 cases, of which the number of deaths is up to 15,660 cases.

Besides social distancing, masking, and handwashing, vaccine is one of the most efficient ways to prevent COVID-19. Most of the vaccines currently available only provide one precursor or vector of protein S, the anti-nucleocapsid (anti-N) antibodies are not fully developed and only anti-S antibodies could be detected (which target spike protein sub-domains, S1 and RBD). On the other hand, due to the biological role of nucleocapsid and the fact that it is protected from antibodies by viral or cellular membranes, nucleocapsid protein (NP) antibodies are unlikely to directly neutralize SARS-CoV-2. For the above-mentioned reasons, screening for anti-S or anti-RBD antibodies is commonly used to investigate the presence of humoral immune markers following a Covid infection or after vaccination.

In the event of vaccination, the duration of antibody persistence is yet unknown. Large cohort studies showed that 90-99% of individuals infected with the SARS-CoV-2 virus developed detectable neutralizing antibodies within 2-4 weeks following infection and immune responses remain robust and protective against reinfection for at least 6-8 months later. In Vietnam, studies on antibody levels after exposure to SARS-CoV-2 or after vaccination are receiving more and more attention. Mai et al. conducted a study to assess the kinetics of antibody titers of eleven COVID-19 infected individuals and found out that the titers of RBD-targeting NAbs decayed by 18-30 weeks after the infection. Chau et al (2021) investigated the vaccine-induced production of neutralizing antibodies after injecting ChAdOx1 nCoV-19 AZD1222 vaccine (Oxford-AstraZeneca) on 554 Vietnamese healthcare workers. This study demonstrated that the concentration of neutralizing antibodies increased after each dose. However, three months after the first dose, neutralizing antibody levels reduced significantly, while the seroconversion rate slightly declined from 98.1% to 94.7% at day 14 after the second dose, but this study did not report neutralizing antibody levels.

Some studies indicated that the efficacy of the Covid-19 vaccine might decrease over time, as demonstrated by the decline of blood antibodies level, thus suggest providing additional booster dose in the hope of increasing protection. However, more information about antibody titers after vaccination is still needed, especially for the Vietnamese population. Therefore, This study is conducted to evaluate the immune response created by the ChAdOx1 nCoV-19 vaccination by measuring the titers of antibodies against the SARS-CoV-2 spike protein receptor binding domain (RBD) among healthcare workers of My Duc Hospital and to investigate potential associations of vaccine protection and infection in this population.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Being vaccinated with at least one dose of ChAdOx1 nCoV-19
* Accepted to take part in the study

Exclusion Criteria:

* Currently being diagnosed with Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare workers of My Duc hospital who were vaccinated with at least one dose of ChAdOx1 nCoV-19.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 anti-RBD IgG concentration | Up to 1 week after examination
  SARS-CoV-2 anti-RBD IgG antibody concentration was reported after analysing the specimen

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — HOPE Research Center, My Duc Hospital
Locations (1):
- HOPE Research Center, My Duc Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No